CLINICAL TRIAL: NCT05989542
Title: An Open, Multi-center, Single-arm Phase IIIb Confirmatory Clinical Study to Evaluate the Efficacy, Safety and Tolerability of Vebreltinib in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer With MET Exon 14 Mutation
Brief Title: A Confirmatory Clinical Study in NSCLC Patients With MET Exon 14 Mutation (KUNPENG-2)
Acronym: KUNPENG-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Pearl Biotechnology Limited Liability Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLB1001-IIIb-NSCLC-01
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PLB1001 (Experimental): Subjects will receive 200mg of PLB1001 twice daily in cycles of 28-day duration until disease progression, death, adverse event (AE) leading to discontinuation or withdrawal of consent.
  Interventions: Drug: PLB1001

INTERVENTIONS:
Drug: PLB1001 — 200mg BID Oral

SUMMARY:
The goal of this clinical trial is to test if PLB1001 works well and safely in Non-small cell lung cancer patients with MET exon 14 mutation. The main questions it aims to answer are:

* If it is works well in Non-small cell lung cancer patients with MET exon 14 mutation
* If it is safety and tolerant in Non-small cell lung cancer patients with MET exon 14 mutation

Participants will

1. be given PLB1001 200mg BID,oral.
2. be received hematology and urine and ECG examinations every 14 days (First 3 months) or every 28 days (After 3 months)
3. be received Image examination every 8 weeks(First year) or every 12 weeks(After one year)

ELIGIBILITY:
Inclusion Criteria:

1. voluntarily sign a written informed consent to participate in the study and be willing and able to comply with study-related visits and procedures;
2. Male or female aged 18 years and above;
3. patients with histologically or cytologically confirmed locally advanced or metastatic non-small cell lung cancer (including sarcomatoid carcinoma of the lung, according to the AJCC 8th edition of lung cancer staging, Stage IIIB - Stage IV) (non-site pathology reports are acceptable);Patients have not received any prior systemic antineoplastic drug therapy for advanced diseaseor disease progression or toxicity intolerance after prior systemic therapy (≤3 lines);
4. The presence of MET exon 14 jump mutation was confirmed by the NGS test in the central laboratory, and the 'Combined Human 9 Gene Mutation Detection Kit (Reversible End Termination Sequencing)' produced by Guangzhou Burning Stone Medical Laboratory Ltd. will be used for the testing and analysis of the samples in the central laboratory. Patients are required to provide sufficient blood samples for retrospective analysis by the central laboratory ('Human Circulating Tumour DNA Multi-Gene Mutation Test Kit (Reversible End Termination Sequencing Method)' manufactured by Guangzhou Burnstone Medical Laboratory Co. Ltd. to support the development of blood companion diagnostic reagents required for the marketing of Piratinib. Note: For patients who have received previous systemic anti-tumour therapy, tumour tissue obtained after disease progression on the most recent anti-tumour therapy will be preferred for biomarker testing;
5. Tissue sample testing confirms EGFR wild-type, ALK rearrangement negative, ROS1 rearrangement negative, and KRAS mutation negative;
6. at least one measurable lesion (per RECIST 1.1 criteria). For a lesion that has received prior radiotherapy, it may be counted as a target lesion only if definitive disease progression has occurred since radiotherapy;
7. an ECOG performance status score of 0-1;
8. expected survival ≥ 3 months;
9. Laboratory tests that meet the following requirements:

   * Aspartate aminotransferase (AST): ≤ 3 x ULN (no liver metastases)
   * Alanine aminotransferase (ALT): ≤3 × ULN (no liver metastases)
   * Total bilirubin (TBIL): ≤1.5 × ULN (no liver metastases)
   * AST: ≤5.0 × ULN (with liver metastases)
   * ALT: ≤5.0 × ULN (with liver metastasis)
   * Total bilirubin: ≤3.0 × ULN (with liver metastases)
   * Platelet count: ≥75 × 10⁹/L (without blood transfusion or mono-collected platelet transfusion or growth factor use within 10 days prior to the start of treatment)
   * Absolute neutrophil count: ≥ 1.5 × 10⁹/L (in the absence of growth factors within 10 days prior to the start of treatment)
   * Hemoglobin > 90 g/L (in the absence of blood transfusion or use of growth factors within 10 days prior to the start of treatment)
   * Coagulation index: INR≤2.0
   * Creatinine clearance (Ccr) >50 mL/min, with Ccr using the Cockcroft-Gault formula: (140 - age[yr]) × body weight (kg) × 1.23 × (0.85, if female)/serum creatinine (μmol/L)
   * Urea/urea nitrogen: ≤1.5 × ULN
   * Asymptomatic serum amylase ≤ grade 2 (NCI-CTCAE 5.0). For patients with Grade 2 serum amylase abnormalities prior to first dose, it is important to confirm that there are no signs and/or symptoms suggestive of pancreatitis or pancreatic injury (e.g., elevated P-amylase, abnormal pancreatic imaging results, etc.)
   * Serum lipase ≤ 1.5 × ULN;
10. the investigator is judged to be compliant and able to complete scheduled visits, treatments and laboratory tests according to the protocol;
11. men and women of childbearing potential must agree to use effective contraception from the time of signing the informed consent until 3 months after the last dose of study drug. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose of study drug.

Exclusion Criteria:

1. unwilling to provide tumor tissue or blood samples for molecular testing;
2. previous treatment with MET inhibitors or HGF-targeted therapy;
3. have symptomatic and neurologically unstable central nervous system (CNS) metastases or CNS disease that requires increased steroid doses for control; NOTE: Patients with CNS metastases whose symptoms have been controlled may be enrolled in this trial. Patients with symptomatic or unstable CNS metastases must have completed radiotherapy, or at least 2 weeks after surgical treatment of CNS tumor metastases, prior to study entry. Patients must have stable neurologic function with no new neurologic deficits identified on clinical examination and no new problems identified on CNS imaging. If the patient requires steroids for the treatment of CNS metastases, they must have been stabilized on a therapeutic dose of steroids for at least 2 weeks prior to signing the informed consent form;
4. patients with clinically poorly controlled pleural, abdominal or pericardial effusions who, in the judgment of the investigator, are not suitable for enrollment;
5. unstable or uncontrolled disease or conditions related to or affecting cardiac function (e.g., unstable angina pectoris, congestive heart failure [NYHA > Class II], unstably controlled hypertension [defined as diastolic blood pressure > 100 mmHg and/or systolic blood pressure > 160 mmHg regardless of antihypertensive medications. initiation of antihypertensive medications or adjustment of antihypertensive medications prior to Screening is permitted]);
6. a coagulation disorder or bleeding tendency, including an arterial or venous thromboembolic event (including myocardial infarction, cerebrovascular accident or transient ischemic attack, pulmonary artery embolism, deep vein thrombosis, or any other history of severe thromboembolism) within 6 months prior to the administration of the first study medication, any life-threatening bleeding event (including the need for transfusional therapy, surgical or topical therapy, and ongoing drug therapy) that Tendency to bleed in the judgment of the investigator;
7. The presence of risk factors for QTc interval prolongation such as chronic hypokalaemia not corrected by complementary therapies, congenital or familial long QT interval syndrome, family history of unexplained sudden death in a first-degree relative under the age of 40 years, or initiation of Piratinib. Patients with a family history of unexplained sudden death in a first-degree relative younger than 40 years of age, or use of a drug that prolongs the QT interval and results in tip-twist ventricular tachycardia for ≤5 half-lives prior to the initiation of the first dose of ponatinib should be excluded.

   Patients with ≤5 half-lives of drugs that prolong the QT interval and cause tip-twist ventricular tachycardia prior to initiation of Brentinib should be excluded.
8. any significant rhythm abnormality such as complete left bundle branch block, second or third degree heart block, medically uncontrolled ventricular arrhythmias, supraventricular, nodal arrhythmias, and medically uncontrolled other cardiac arrhythmias;
9. active gastrointestinal disorders (e.g., ulcerative lesions, uncontrollable nausea, vomiting, diarrhea, and malabsorption syndromes) or other conditions (e.g., inability to swallow the test medication, or prior major gastrointestinal surgery) that significantly interfere with absorption, distribution, metabolism, or excretion of the oral study drug;
10. the presence of an active infection, including but not limited to: 1) Hepatitis B (Hepatitis B Surface Antigen [HBsAg] positive and Hepatitis B Virus [HBV] DNA ≥ 500 IU/ml), Hepatitis C (positive for both anti-Hepatitis C Virus [HCV] antibodies and HCV-RNA) or Human Immunodeficiency Virus (HIV) (HIV antibody positive) infections, and syphilis positive infections; 2) Active tuberculosis; 3) Active infection (e.g., pneumonia) requiring systemic anti-infective therapy within 2 weeks prior to first study drug administration;
11. known history of hypersensitivity to the active or inactive excipients of Vebreltinib, hypersensitivity to drugs with a chemical structure similar to that of Vebreltinib.
12. patients being treated with warfarin or any other coumarin derivative anticoagulant, with the exception of low-dose warfarin (< 2 mg) for the prevention of central catheter-related thrombosis;
13. presence of prior antineoplastic therapy toxicity not recovered to ≤ Grade 1 (NCI-CTCAE 5.0) or baseline, except for alopecia, skin hyperpigmentation, and Grade 2 peripheral neurotoxicity
14. any comorbid medical condition that may increase the risk of toxicity;
15. antineoplastic and investigational drug therapy within 2 weeks or ≤ 5 drug half-lives (whichever is longer, up to a maximum of 4 weeks) prior to initiation of the first dose of Vebreltinib. If the prior therapy was a monoclonal antibody, the therapy must be discontinued at least 2 weeks prior to the first dose of Vebreltinib. If the prior therapy was an oral targeted drug, the therapy must be discontinued at least 5 drug half-lives (up to 4 weeks) prior to the first dose of Vebreltinib. If prior therapy was an herbal antineoplastic therapy, it must be discontinued at least 1 week prior to the first dose of Vebreltinib;
16. chest radiotherapy to the lung field ≤ 4 weeks prior to initiating treatment with Vebreltinib or if the patient has not recovered to ≤ Grade 1 from radiotherapy-related toxicity. For all other sites (including radiotherapy to the thoracic spine or ribs), radiotherapy ≤ 2 weeks prior to initiation of Vebreltinib therapy or the patient has not recovered from radiotherapy-related toxicity. Palliative radiotherapy to bone metastatic lesions for pain relief does not require a washout period;
17. major surgery (e.g., intrathoracic, intra-abdominal, or intra-pelvic) within 4 weeks prior to initiation of treatment with Vebreltinib, brain metastasectomy may be relaxed to within 2 weeks or if the patient has not recovered from the side effects of these surgeries or is significantly traumatized, or if the patient is expected to have a significant surgical need during the study period. Thoracoscopic biopsy procedures and mediastinoscopy are not considered major surgery and patients may be enrolled ≥1 week after the procedure;
18. another malignancy diagnosed within the last 3 years in addition to NSCLC and/or requiring treatment. Completely resected basal cell and squamous skin cancers, and completely resected carcinoma in situ of any type are excluded;
19. patients are treated with CYP3A4 potent inducer and/or potent inhibitor medications that cannot be discontinued for at least 1 week prior to initiation of treatment with Vebreltinib and for the duration of the study;
20. is pregnant or is breastfeeding
21. is currently participating in another interventional clinical trial or has received an investigational drug within 2 weeks prior to the first dose of the test drug
22. other circumstances that, in the opinion of the investigator, make participation in the study inappropriate, such as the presence of evidence of severe or uncontrolled systemic disease, including, but not limited to, active primary immunodeficiency disease, allogeneic organ transplantation, that make the patient unsuitable for participation in this trial or that would impede adherence to the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Confirmed Objective Response Rate Evaluated by IRC | 2 years
  Objective response rate will be determined according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Objective response rate is defined as the percentage of patients who experienced either a complete response (CR) or partial response (PR) from first administration of trial treatment to first observation of progressive disease (PD). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30 percent (%) reduction from baseline in the sum of the longest diameter (SLD) of all lesions. PD is defined as at least a 20% increase in the SLD, but at least increase 5mm, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.

SECONDARY OUTCOMES:
Confirmed Objective Response Rate evaluated by Investigator | 2 years
  Objective response rate will be determined according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Objective response rate is defined as the percentage of patients who experienced either a complete response (CR) or partial response (PR) from first administration of trial treatment to first observation of progressive disease (PD). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30 percent (%) reduction from baseline in the sum of the longest diameter (SLD) of all lesions. PD is defined as at least a 20% increase in the SLD, but at least increase 5mm,taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Disease Control Rate evaluated by IRC and Investigator | 2 years
  Disease Control Rate according to RECIST 1.1 is the percentage of patients who experienced either a complete response (CR), partial response (PR) or stable disease (SD).
Duration Of Response evaluated by IRC and Investigator | 2 years
  Duration Of Response according to RECIST 1.1 is the time from when the CR/PR (whichever is first) criteria are first met until progression of disease (PD) or death due to any cause.
Time To Response evaluated by IRC and Investigator | 2 years
  Time To Response according to RECIST 1.1 is the time from the first trial treatment administration to the CR/PR (whichever is first) criteria are first met.
Progression Free Survival evaluated by IRC and Investigator | 2 years
  Progression Free Survival is defined as the time (in months) from the first administration of trial treatment to the date of the first documentation of PD or death due to any cause.
Intracranial Duration Of Response evaluated by IRC and Investigator | 2 years
  Duration Of Response according to RECIST 1.1 is the time from when the CR/PR (whichever is first) criteria are first met until progression of disease (PD) or death due to any cause.
Intracranial Disease Control Rate evaluated by IRC and Investigator | 2 years
  Disease Control Rate according to RECIST 1.1 is the percentage of patients who experienced either a complete response (CR), partial response (PR) or stable disease (SD).
Intracranial Time To Response evaluated by IRC and Investigator | 2 years
  Time To Response according to RECIST 1.1 is the time from the first trial treatment administration to the CR/PR (whichever is first) criteria are first met.
Intracranial Progression Free Survival evaluated by IRC and Investigator | 2 years
  Progression Free Survival is defined as the time (in months) from the first administration of trial treatment to the date of the first documentation of PD or death due to any cause.
Occurrence of Treatment emergent adverse event (TEAEs) | 2 years
  This outcome measure will be presented as the percentage of subjects with any (serious) adverse event (AE). Percentages are calculated using total number of subjects per treatment cohort as the denominator.

OTHER OUTCOMES:
Minimum plasma concentration (Cmin) of drug and safety-analysis-set.etc | Within 2 hours prior to morning dose on day 1 (±7) of Cycle 2,Cycle,3,Cycle5 (eash cycle is 28 days )
  Subjects need collect PK sample within 2 hours prior to morning dose on day 1 (±7 days) of cycles 2, 3, and 5.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No